CLINICAL TRIAL: NCT04089267
Title: Multicenter, Randomized, Open, Parallel Controlled Trials Evaluating the Efficacy and Safety of Different Human Thrombopoietin (rhTPO) Regimens in the Treatment of Patients With Primary Immune Thrombocytopenia (ITP)
Brief Title: Evaluating the Efficacy and Safety of Different Human Thrombopoietin (rhTPO) Regimens in the Treatment of Patients With Primary Immune Thrombocytopenia (ITP)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shenyang Sunshine Pharmaceutical Co., LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3sbio-TPO-403
Record Dates: First submitted 2019-09-10; First posted 2019-09-13 (Actual); Last update posted 2019-09-13 (Actual); Status verified 2019-09

CONDITIONS: ITP

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- experimental group 1 (Experimental): rhTPO injection7500 U ;one time a day; 14 times of administration
  Interventions: Drug: TPO
- experimental group 2 (Experimental): rhTPO injection15000 U;one time a day;14 times of administration
  Interventions: Drug: TPO
- experimental group 3 (Experimental): rhTPO injection15000 U;1 time every other day, 7 times;
  Interventions: Drug: TPO
- experimental group 4 (Experimental): rhTPO injection30000 U；1 time every other day, 7 times;
  Interventions: Drug: TPO

INTERVENTIONS:
Drug: TPO

SUMMARY:
This is a review of the efficacy and safety of different recombinant human thrombopoietin (rhTPO) regimens in the treatment of patients with primary immune thrombocytopenia (ITP).

DETAILED DESCRIPTION:
Evaluating the efficacy and safety of different human thrombopoietin (rhTPO) regimens in the treatment of patients with primary immune thrombocytopenia (ITP) This trial was designed as a multicenter, randomized, open, parallel controlled study

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old, male or female
* For patients who have been diagnosed with ITP, the diagnostic criteria are consistent with the Chinese Expert Consensus on Diagnosis and Treatment of Primary Immune Thrombocytopenia (2016 Edition)
* Recurrence after previous treatment with glucocorticoids is ineffective or effective
* No contraindications to rhTPO (Terbyus) application, and willing to accept rhTPO treatment
* Platelet count before enrollment ≤ 30 × 109 / L, or > 30 × 109 / L but with active bleeding
* Volunteer to participate in the study and sign the informed consent form

Exclusion Criteria:

* pregnant or lactating
* Those with a history of thrombosis
* severe cardiopulmonary liver and kidney dysfunction: creatinine level ≥ 176.8μmol / l (2mg / dl), transaminase, bilirubin levels higher than the upper limit of the normal value of 3 times
* Those who have used rhTPO in the past 2 weeks, or who have undergone splenectomy within 2 months, or who have been treated with danazol for less than 1 month, or have recently applied the following ITP treatments but have not yet reached the efficacy judgment time. : C-ball (7 days), vincristine or vinblastine amide or rhIL-11 (2 weeks), Eltrombopag (1 month), or rituximab (2 months)
* In the case of previous treatment of rhTPO: rhTPO 300U/kg/d, 14 days of treatment is invalid;
* Severe or uncontrollable infections
* have a history of mental illness
* The investigator believes that the patient is not eligible to participate in any other circumstances of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
The change in Platelet count from baseline on day 14 after the first dose | for day 14
Total effective rate of ITP patients on day 14 (V6, D14 ± 1) after the first dose. | for day 14

SECONDARY OUTCOMES:
The change in Platelet count from baseline on day 7 and day28 after the first dose | for day7and day28
the total effective rate of treatment in ITP patients on day 7 and day 28 | for day7and day28
AE | up to 28days
Incidence of anti-rhTPO antibodies | up to 28days
Cav | up to 28days
  average Blood concentration at steady state Blood concentration at steady state Blood concentration at steady state
AUCss | up to 28days

CONTACTS AND LOCATIONS:
Locations (21):
- China (21):
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Zhongshan Hospital Xiamen University, Xiamen, Fujian
  - The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Guangdong Second People's Hospital, Guangzhou, Guangdong
  - Guangzhou Panyu Central Hospital, Guangzhou, Guangdong
  - Harbin Institute of Hematology and Oncology, Haerbin, Heilongjiang
  - Henan University of Science and Technology First Affiliated Hospital, Luoyang, Henan
  - The First Affiliated Hospital of Henan University of Traditional Chinese Medicine, Zhengzhou, Henan
  - Zhengzhou Central Hospital, Zhengzhou, Henan
  - renmin Hospital of Wuhan University Hubei General Hospital, Wuhan, Hubei
  - Loudi Central Hospital, Loudi, Hunan
  - The Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - First Affiliated Hospital Heilongjiang University of Chinese Medicine, Shenyang, Liaoning
  - Xi An Central Hospital, Xi’an, Shanxi
  - Chinese Academy of Medical Sciences Blood Disease Hospital, Tianjin, Tianjin Municipality
  - Xinjiang Uygur Autonomous Region Chinese Medicine Hospital,, Ürümqi, Xinjiang
  - Affiliated Hangzhou First People's Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Lishui City Center Hospital, Lishui, Zhejiang
  - The First Affiliated Hospital of Xinjiang Medical University, Xinjiang
  - Xinxiang Central Hospital,, Xinxiang

IPD SHARING:
Plan to Share IPD: Yes